CLINICAL TRIAL: NCT02708199
Title: Molecular Assessment of Drug Resistance Markers in Asymptomatic Malaria Cases in Myanmar Artemisinin Resistance Containment Zones and Malaria Antibody Kinetic Analysis
Brief Title: Molecular Assessment of Drug Resistance Markers in Asymptomatic Malaria Cases and Malaria Antibody Kinetic
Status: Completed | Type: Observational
Sponsor: Department of Medical Research, Lower Myanmar (Other)
Collaborators: Kangwon National University (Other)
Responsible Party: Principal Investigator, Myat Htut Nyunt, Research Scientist, Department of Medical Research, Lower Myanmar
Other Study IDs: KMRL_01_2016
Record Dates: First submitted 2016-03-05; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Increased Drug Resistance; Asymptomatic Infection; Malaria
Keywords: Drug resistance malaria; Myanmar Artemisinin Resistance Containment Zone; Asymptomatic malaria; Serology
MeSH Terms: conditions — Asymptomatic Infections; Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples have been collected and DNA have been extracted and keep at -20 degree C until analysis. Sera were also separately keep at -80 degree C until analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
Detection of the drug resistance molecular markers for falciparum and vivax in Longitudinal follow-up samples collected in Shwegyin Township, Bago Region that is Artemisinin Resistance Containment Tier I.

DETAILED DESCRIPTION:
This study is longitudinal and observational cohort study to detect the drug resistance molecular markers in asymptomatic malaria infected local residents in study site. Only local residence who are not migrants, are recruited in the study and active and passive surveillance have been carried out within one year observation period. At the time of enrollment, blood film examination, rapid diagnosis test (RDT) testing have been done all together with the collection of the venous blood (about 1-2 mL) that would be used for molecular analysis later. All of the RDT or microscopy positive cases were treated according to the National Malaria Treatment Policy in Myanmar. A total of at least 1000 participants have been recruited in the study. Active case detection has been done in every three months. The venous blood were used for molecular based detection of the asymptomatic malaria infection by using High-throughout pooling strategy. All of the positive samples, (falciparum and vivax), have been checked for drug resistance molecular analaysis compared with the previously collected symptomatic malaria infection cases in the same region.

ELIGIBILITY:
Inclusion Criteria:

* Local resident in stud sites
* Who give informed consent
* No known tentative plan to move/ migrant elsewhere within one year

Exclusion Criteria:

* Migrant or mobile population
* Less than 6 year

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Shwegyin Township, Bago Region, Myanmar Artemisinin resistance containment Zone I.
Sampling Method: Non-Probability Sample
Enrollment: 1179 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of the Asymptomatic malaria infection | 2016 March
  Number of the asymptomatic malaria infection by molecular method in the sample collected from apparently healthy individuals. It have been done by nested PCR based method. Number of the asymptomatic infection will be finished in March 2016. (up to up to 5 months after last samples collection)

SECONDARY OUTCOMES:
Number of the cases that showed drug resistance molecular markers in asymptomatic malaria infection | 2016 April
  K13, Pffd, Pfmdr2 and Pfcrt markers for falciparum and Pvcrt-O, Pvdhps, Pvdhfr and Pvmdr1 for vivax asymptomatic infections.The target sequences will be analysed to detect the specific single nucleotide polymorphism (SNPs). Molecular marker analysis will be done as soon as after asymptomatic infection have been confirmed. It will be finished in 2016 April. (up to 6 months after last sample collection)
Prevalence of the different Malaria Antibody in local resident in Myanmar | 2016 December
  Malaria antibody that against the malaria parasites will be assessed by using high sensitive protein microarray. Total overall prevalence will be assessed and time to time change of the antibody status will be observed. It will be started in April until December 2016.(Up to 14 months after last sample collection)

IPD SHARING:
Plan to Share IPD: Undecided
The data may be shared after publish.